CLINICAL TRIAL: NCT01925898
Title: A Randomized, Clinical Trial of Oral Midazolam Versus Oral Ketamine for Sedation During Laceration Repair.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 87/13
Record Dates: First submitted 2013-07-17; First posted 2013-08-20 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2013-08

CONDITIONS: Lacerations
Keywords: Laceration; Sedation; Pediatrics
MeSH Terms: conditions — Lacerations | interventions — Midazolam; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ketamine (Experimental): Oral ketamine
  Interventions: Drug: Experimental Arm: Ketamine
- Midazolam (Active Comparator): Oral Midazolam
  Interventions: Drug: Midazolam - active comparator

INTERVENTIONS:
Drug: Midazolam - active comparator — Oral midazolam - 0.7mg/kg single dose
  Other Names: Dormicum
  Arms: Midazolam
Drug: Experimental Arm: Ketamine — Oral Ketamine 5mg/kg Single dose
  Other Names: Ketalar
  Arms: Ketamine

SUMMARY:
Sedation is often needed for young children undergoing minor procedures in the emergency department (ED). Oral midazolam is one of the most commonly used regimens for children undergoing laceration repair but its sedative efficacy was shown to be suboptimal. In only one randomized controlled study oral ketamine has been used successfully for procedural sedation for laceration repair. A recent study showed that the combination of oral midazolam and oral ketamine provided deeper sedation compared with oral midazolam alone. However children treated wuth the combination of midazolam and ketamine required longer recovery

Hypothesis:

Oral ketamine can provide superior sedation to oral midazolam in children requiring sedation for laceration repair.

ELIGIBILITY:
Inclusion Criteria:

• Any child with laceration requiring sedation

Exclusion Criteria:

* Major trauma
* Closed head injury associated with loss of consciousness
* Abnormal neurologic examination in a previously normal child
* Significant developmental delay or baseline neurological deficit
* A patient with seizures
* Elevated intra-cranial pressure
* Hypersensitivity to midazolam or ketamine
* Hypertension
* Hyperthyroidism or a patient receiving thyroid replacement
* alcohol intoxication or a history of alcohol abuse
* Acute or chronic respiratory, cardiac, renal or hepatic abnormalities
* Glaucoma
* Known psychiatric disease
* American Society of Anesthesiologists (ASA) score of more than 2
* Informed consent cannot be obtained from legal guardian

Ages: 1 Year to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2013-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-07 (Estimated)

PRIMARY OUTCOMES:
Pain score: Visual analog score (VAS)- by a parent | During the procedure - up to 1 hour
  A parent will assess the child's pain on a Visual analog scale
Number of patients requiring IV sedation | During the procedure - up to 1 hour
  patients who fail to achieve University of Michigan Sedation Scale (UMSS) of two or higher will be switched to IV sedation

SECONDARY OUTCOMES:
UMSS - by ED physician | During the procedure - up to 1 hour
• VAS by nurse | During the procedure - up to 1 hour
Time to reach UMSS > 2 | up to 1 hour
• Procedure time | During the procedure - up to 1 hour
• Time from procedure to full recovery | While in the ED - estimated time around 2 hours
The occurrence of adverse effects during the ED stay | While in the ED - estimated time around 2 hours
  Significant adverse effects are defined as
  1. Oxygen desaturation <92% or hypoventilation requiering ventilatory support
  2. Need for hemodynamic support
  3. Anaphylaxis
  4. Seizures
  5. Any adverse effects requiring patient admission
• Patients and parents satisfaction assessed on VAS | While in the ED - estimated time around 2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh MC, Be’er Ya‘aqov, Israel